CLINICAL TRIAL: NCT05107284
Title: Personalized Feedback After Alcohol Health Education for Members of Greek Life (GREEK Study)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Abby Braitman (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Abby Braitman, Assistant Professor, Old Dominion University
Organization: Old Dominion University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-164; K01AA023849 (NIH)
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: College Student Drinking
MeSH Terms: conditions — Alcohol Drinking in College

STUDY DESIGN:
Who Masked: Participant
Masking Description: The intervention is an online program, not an individual administering it, so masking is not necessary. Similarly, the same online survey is deployed in all follow-up assessments regardless of condition, and data are not collected by individuals, so masking of investigators is not necessary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention-only Control (Placebo Comparator): Participants navigate through e-checkup to go, the well-established alcohol intervention. Any follow-up emails sent to them later contain only a reminder to participate in follow-up surveys.
  Interventions: Behavioral: e-checkup to go
- Intervention plus delayed feedback booster (Experimental): Participants navigate through e-checkup to go, the well-established alcohol intervention, then receive a series of feedback booster emails. It contains a reminder to participate in follow-up surveys, plus personalized feedback based on participant-reported perceived alcohol norms, actual alcohol norms, their own use, and harm reduction strategies.
  Interventions: Behavioral: e-checkup to go; Behavioral: Delayed feedback booster

INTERVENTIONS:
Behavioral: e-checkup to go — The e-checkup to go alcohol program is designed to motivate individuals to reduce their alcohol consumption using personalized information about their own use and risk factors. The program is a combination of several components including alcohol education, personalized feedback, attitude-focused strategies, and skills training. It is self-guided and requires no face-to-face time with an administrator. It provides tailored feedback regarding quantity and frequency of alcohol use, normative comparisons, physical health information, amount and percent of income spent on alcohol, negative consequences feedback, explanation and advice for how to reach their goals, and resources.
Behavioral: Delayed feedback booster — Booster emails will contain normative feedback indicating average consumption for students at the same institution by sex, their perceptions of student drinkers at the same institution, their own reported consumption, and reminders of strategies they can use to protect themselves from alcohol-related harm.
  Arms: Intervention plus delayed feedback booster

SUMMARY:
Heavy episodic alcohol use within the college student population is widespread, creating problems for student drinkers, their peers, and their institutions. Negative consequences from heavy alcohol use can be mild (e.g., hangovers, missed classes), to severe (e.g., assault, even death). Although online interventions targeting college student drinking reduce alcohol consumption and associated problems, they are not as effective as in-person interventions. Online interventions are cost-effective, offer privacy, reduce stigma, and may reach individuals who would otherwise not receive treatment. In a recently completed randomized, controlled trial, an emailed booster with personalized feedback improved the efficacy of a popular online intervention. A second randomized, controlled trial confirmed efficacy for students of legal drinking age for a longer timeline. Although promising, the booster incorporated in the study needs further empirical refinement.

The current project seeks to build on past progress by further developing and refining the booster. In particular, the current project is an extension of previous work by expanding the investigation into complete social networks (students involved in Greek life). This booster contains feedback about alcohol use tailored to the recipient, and will be emailed 2, 6, 10, and 14 weeks after baseline (experimental condition), or not at all (control condition). This study will be conducted specifically with students who are members of fraternities or sororities at ODU (specifically, those in the organizations that agree to participate). This population engages in heavy alcohol use so is ideal for an alcohol intervention. Members of fraternities and sororities (i.e., "Greek life") engage in more frequent drinking, consume more when drinking, and have higher peak drinking occasions than students not involved in Greek life. We aim to administer the intervention and associated booster among complete networks of Greek organizations to examine how the intervention and booster and progress through social networks.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years old so that they can legally consent to participate.
* Participants must be an undergraduate student at the host institution and a member of a participating fraternitiy or sorority.

Exclusion Criteria:

* Under 18 years of age
* Not a member of a participating fraternity or sorority at the host institution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Alcohol consumption | past 30 days
  Participant self-reported number of standard drinks consumed by participant over a typical week for the past 30 days.

SECONDARY OUTCOMES:
Alcohol-Related Consequences | past 30 days
  Participant self-report on the Brief-Young Adult Alcohol Consequences Questionnaire (B-YAACQ; Kahler et al., 2005), which assesses alcohol-related problems experienced by the participant. Total scores are created by summing all individual items, and range from 0 to 24, with higher values representing more problems experienced (i.e., worse outcomes).

CONTACTS AND LOCATIONS:
Overall Officials: Abby L Braitman, Ph.D., Principal Investigator — Old Dominion University
Locations (1):
- Old Dominion University, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Braitman AL, Lau-Barraco C. Personalized Boosters After a Computerized Intervention Targeting College Drinking: A Randomized Controlled Trial. Alcohol Clin Exp Res. 2018 Sep;42(9):1735-1747. doi: 10.1111/acer.13815. Epub 2018 Jul 11. PMID 29995326
- [Background] Braitman AL, Henson JM. Personalized boosters for a computerized intervention targeting college drinking: The influence of protective behavioral strategies. J Am Coll Health. 2016 Oct;64(7):509-19. doi: 10.1080/07448481.2016.1185725. Epub 2016 May 5. PMID 27148633
- [Background] Braitman AL, Strowger M, Lau-Barraco C, Shipley JL, Kelley ML, Carey KB. Examining the added value of harm reduction strategies to emailed boosters to extend the effects of online interventions for college drinkers. Psychol Addict Behav. 2022 Sep;36(6):635-647. doi: 10.1037/adb0000755. Epub 2021 Jun 3. PMID 34081487
- [Derived] Braitman AL, Shipley JL, Strowger M, Ayala Guzman R, Whiteside A, Bravo AJ, Carey KB. Examining Emailed Feedback as Boosters After a College Drinking Intervention Among Fraternities and Sororities: Rationale and Protocol for a Remote Controlled Trial (Project Greek). JMIR Res Protoc. 2022 Oct 28;11(10):e42535. doi: 10.2196/42535. PMID 36306162

DOCUMENTS (2):
  • Study Protocol (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/84/NCT05107284/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/84/NCT05107284/SAP_001.pdf